CLINICAL TRIAL: NCT05172089
Title: Diabetic Foot Ulcer (DFU) Biofilm Infection and Recurrence
Acronym: DFUBiofilm
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Arizona (Other)
Responsible Party: Principal Investigator, Chandan Sen, Professor, University of Pittsburgh
Other Study IDs: STUDY23050116; 3R01DK125835-02S1 (NIH)
Record Dates: First submitted 2021-12-12; First posted 2021-12-29 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Chronic Wounds; Biofilm Infection; Trans-epidermal Water Loss (TEWL); Diabetic Foot; Diabetic Foot Infection
Keywords: foot ulcer; diabetic foot; wound infection; diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Wound Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Wound debridement collection: Debridement of tissue will be conducted as a standard of care (SoC) procedure for these patients. This debrided tissue would normally be disposed of as waste tissue, but for this study the investigators will collect this discarded waste tissue and perform analysis. In brief, waste tissue from debridement of the wound edge will be collected for histology molecular biology and immunohistochemistry studies. Samples will be used to determine whether the wound is infected using standard lab techniques.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic Foot Ulcer study: 405 clinically diagnosed Diabetic Foot Ulcer (DFU) patients who are suspected to be infected will be recruited . Wound swab for culture obtained. Baseline digital imaging of target wound(s). SF-12 Health survey, Visual Analogue Pain scale, Cardiff wound impact questionnaires. Wound site evaluation including TcOM/TBI/ankle brachial index (ABI) will be completed for subjects with wounds below the knee, if not already completed per standard of care within the previous 12 months. Hemoglobin A1c point of care testing will be drawn for diabetic subjects who do not have an A1c available within 90 days prior to enrollment; 3mm biopsy tissue or debrided tissue will be collected. Ideally, two tissue samples will be obtained; the subject's medical records will be reviewed and followed for up to 16 weeks or until their wound has closed, whichever comes first. The research staff will also call the patient or care facility as needed to check for wound closure.

SUMMARY:
This work is based on DFU patients, seeks to conduct a fully powered clinical study testing i) If DFU with a history of biofilm infection closes with deficient barrier function. ii) whether such functionally deficient wound closure, manifested as high TEWL, is associated with greater wound recurrence. The primary parent study will also address molecular mechanisms implicated in biofilm-induced loss of skin epithelial barrier integrity in DFU patients.

DETAILED DESCRIPTION:
Diabetic foot ulcers (DFU) are one of the most common reasons for hospitalization of diabetic patients and frequently results in amputation of lower limbs. Of the one million people who undergo non-traumatic leg amputations annually worldwide, 75% are performed on people who have type 2 diabetes (T2DM). The risk of death at 10 years for a diabetic with DFU is twice as high as the risk for a patient without a DFU. The rate of amputation in patients with DFU is 38.4%4. Infection is a common (>50%) complication of DFU. Emerging evidence underscores the significant risk that biofilm infection poses to the non-healing DFU. Biofilms are estimated to account for 60% of chronic wound infections. In the biofilm form, bacteria are in a dormant metabolic state. Thus, standard clinical techniques like the colony forming unit (CFU) assay to detect infection may not detect biofilm infection. Thus, biofilm infection may be viewed as a silent maleficent threat in wound care.

n the current standard of care (SoC), wound closure is defined (FDA) by wound area re-epithelialization without drainage. The investigators' pre-clinical large animal work demonstrates that wounds with a history of biofilm infection may meet above criteria, but the repaired wound-site skin is deficient in barrier function. This has led to the concept of functional wound closure wherein the current clinical definition of wound closure is supplemented with a functional parameter - restoration of skin barrier function as measured by low trans-epidermal water loss (TEWL).

This study rests pilot study showing that closed DFU with deficient barrier function are more likely to recur. Biofilm infection as assessed through scanning electron microscopy and wheat germ agglutin assay performed on debrided tissue causes faulty re-epithelialization, compromising skin barrier function at the closed wound site. This work is based on DFU patients, seeks to conduct a fully powered clinical study testing i) If DFU with a history of biofilm infection closes with deficient barrier function. ii) whether such functionally deficient wound closure, manifested as high TEWL, is associated with greater wound recurrence. The primary parent study will also address molecular mechanisms implicated in biofilm-induced loss of skin epithelial barrier integrity in DFU patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, Age ≥ 18
* Willing to comply with protocol instructions, including all study visits and study activities.
* Patient with an open Diabetic Foot Ulcer
* Adequate arterial blood flow as evidenced by at least one of the following (for wounds below the knee):
* TcOM >30 mmHg
* Ankle-brachial index ≥0.7-1.20
* Toe pressure > 30 mmHg
* TBI > 0.6 mmHg

Exclusion Criteria:

* Individuals who are deemed unable to understand the procedures, risks, and benefits of the study.
* Wounds closed or to be surgically closed by flap or graft coverage
* Subjects with marked immunodeficiency (HIV/AIDS, or on immunosuppressive medications.
* TcOM < 30mmHg
* Diabetics with a hemoglobin A1c > 12 within 3 months prior to enrollment
* Subject with autoimmune connective tissue disease
* Ulcer size and location that does not allow the TEWL measurement per SOP
* Pregnant women
* Prisoners
* Unable to comply with study procedures and/or complete study visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinically diagnosed Diabetic Foot Ulcer (DFU) patients who are suspected to be infected will be recruited for this larger cohort of patients in the parent study.
Sampling Method: Probability Sample
Enrollment: 405 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2028-06-27 (Estimated); Study Completion 2029-06-27 (Estimated)

PRIMARY OUTCOMES:
Biofilm infection abundance | 16 weeks
  Test the incidence of wound biofilm infection at initial visit and test its association with deficient skin barrier function at the closed DFU-site
TEWL | 12 weeks
  Trans epidermal water loss post closure and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chandan K Sen, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - UPMC Wound Healing Services at UPMC Passavant, Cranberry Township, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT05172089/ICF_000.pdf